CLINICAL TRIAL: NCT01987843
Title: A Phase IIa, Multicentre, Randomised, Double-Blind, Parallel Group, Placebo-Controlled Study to Evaluate Safety, Tolerability and Clinical Efficacy of MT-1303 in Subjects With Moderate to Severe Chronic Plaque Psoriasis
Brief Title: Dose-finding Study of MT-1303 in Subjects With Moderate to Severe Chronic Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MT-1303-E06
Record Dates: First submitted 2013-11-13; First posted 2013-11-19 (Estimated); Last update posted 2014-12-18 (Estimated); Status verified 2014-12

CONDITIONS: Plaque Psoriasis
Keywords: Psoriasis; Plaque Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- MT-1303-Low (Experimental): MT-1303-Low Dose
  Interventions: Drug: MT-1303-Low
- MT-1303-Middle (Experimental): MT-1303-Middle Dose
  Interventions: Drug: MT-1303-Middle
- MT-1303-High (Experimental): MT-1303-High Dose
  Interventions: Drug: MT-1303-High
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MT-1303-Low
  Arms: MT-1303-Low
Drug: MT-1303-Middle
  Arms: MT-1303-Middle
Drug: MT-1303-High
  Arms: MT-1303-High
Drug: Placebo
  Arms: Placebo

SUMMARY:
The primary objectives of the study are:

* To evaluate the safety and tolerability of three dose levels of MT-1303 in subjects with moderate to severe chronic plaque psoriasis.
* To evaluate the efficacy of three doses levels of MT-1303 in subjects with moderate to severe chronic plaque psoriasis compared to placebo after 16 weeks of treatment on Psoriasis Area and Severity Index (PASI).

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed with plaque psoriasis for at least 6 months prior to screening
* Have moderate to severe chronic plaque psoriasis as defined by PASI score ≥ 12 and BSA ≥ 10% at baseline
* In the investigator's opinion is a candidate for systemic therapy

Exclusion Criteria:

* Non-plaque forms of psoriasis (e.g., guttate, erythrodermic or pustular)
* Current drug-induced or aggravated psoriasis (e.g., a new onset of psoriasis or an exacerbation of psoriasis from beta-blockers, calcium-channel blockers, or lithium carbonate)
* History of any of a list of pre-defined cardiovascular diseases
* History or known presence of any significant infectious, metabolic, oncological, ophthalmological or respiratory system disease or illness likely to render the subject unsuitable for the study.
* Previous exposure to any other S1P receptor modulator
* Receipt of a live vaccine within 28 days prior to randomisation
* Need, or likely need for, treatment with Class I or III anti-arrhythmic drugs or with heart-rate-lowering beta-blockers or calcium-channel blockers, or with any other drugs which can reduce the heart rate
* Clinically significant findings electrocardiogram (ECG) findings.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2013-09; Primary Completion 2014-09 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who achieve PASI 75 (at least 75% reduction from baseline) | 16 weeks

CONTACTS AND LOCATIONS:
Locations (52):
- Bulgaria (3):
  - Research Site, Dupnitsa
  - Research Site, Pleven
  - Research Site, Sofia
- Estonia (2):
  - Research Site, Tallinn
  - Research Site, Tartu
- Germany (11):
  - Research Site, Bavaria
  - Research Site, Cologne
  - Research Site, Düsseldorf
  - Research Site, Essen
  - Research Site, Gera
  - Research Site, Hamburg
  - Research Site, Hanau
  - Research Site, Hessen
  - Research Site, Kiel
  - Research Site, Lübeck
  - Research Site, Mainz
- Hungary (5):
  - Research Site, Debrecen
  - Research Site, NyÃ-regyhÃ¡za
  - Research Site, Orosháza
  - Research Site, Szeged
  - Research Site, Veszprém
- Latvia (4):
  - Research Site, Jelgava
  - Research Site, Madona
  - Research Site, Riga
  - Research Site, Ventspils
- Poland (11):
  - Research Site, Bialystok
  - Research Site, Bydgoszcz
  - Research Site, Gdansk
  - Research Site, Katowice
  - Research Site, Lodzkie
  - Research Site, Malopolska
  - Research Site, Olsztyn
  - Research Site, Środa Wielkopolska
  - Research Site, Warsaw
  - Research Site, Woj. Wielkopolskie
  - Research Site, Wroclaw
- Russia (5):
  - Research Site, Chelyabinsk
  - Research Site, Moscow
  - Research Site, Saint Petersburg
  - Research Site, Saratovskaya
  - Research Site, Yaroslavl
- Ukraine (11):
  - Research Site, Dniepropetrovsk
  - Research Site, Dnipro
  - Research Site, Donetskaya
  - Research Site, Kyiv
  - Research Site, Luhansk
  - Research Site, Lviv
  - Research Site, Odesa
  - Research Site, Simferopol
  - Research Site, Ternopil
  - Research Site, Uzhhorod
  - Research Site, Zaporizhzhya